CLINICAL TRIAL: NCT01111786
Title: Durometer Skin Assessment in Scleroderma: a Study to Validate This New Tool in the Digital Tufts
Brief Title: Finger Hardness Measure in Scleroderma
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Thomas Osborn, MD, Mayo Clinic
Other Study IDs: 09-007486
Record Dates: First submitted 2010-04-05; First posted 2010-04-28 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Scleroderma
Keywords: scleroderma; skin; tightness; durometer
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Thirty subjects with systemic sclerosis and 30 age and sex matched controls without any known condition that should cause increased skin hardness in the fingers with undergo examination by manual palpation and durometer measured hardness of their digital tuft skin by 2 observers on 2 separate occasions. There will be 1 hour between individual observer's scorings. Observers will be blinded from the observer's scores and from their previous scores. Results will be tabulated and compared for manual scores versus durometer measurements, intra-observer scores by both methods and inter-observer scores by both methods.

DETAILED DESCRIPTION:
It is pretty straightforward. We will measure and record the hardness of the digital tufts on ten digits by palpation and the hardness in the same area by using a durometer. We will repeat this one hour later. Scores will be compared as a measure of how consistent and precise they are.

ELIGIBILITY:
Inclusion Criteria:

* Scleroderm
* Rheumatologic condition not effecting the skin tightness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Scleroderma and controls without tight skin attending our rheumatology clinic for a regularly schedualled visit
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Fingertip hardness in patients with scleroderma and controls: comparing manual assessment(scale0 - 3) with durometer assessment(scale 0- 100). | 1 year
  Two investigators will compare data from 30 patients with scleroderma and 30 control patients without fingertip inflammation or tightness twice using durometer readings to those done by manual palpation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Osborn, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States